CLINICAL TRIAL: NCT02102607
Title: Effect of Age on the Median Effective Dose(ED50) for Motor Block With Intrathecal Ropivacaine
Acronym: Spinal
Status: Completed | Type: Observational
Sponsor: China Three Gorges University, Yichang, China (Other)
Responsible Party: Principal Investigator, Mingquan Chen, the First College of Clinical Medical Science, China Three Gorges University (China), China Three Gorges University, Yichang, China
Other Study IDs: intrathecal ropivacaine; China Three Gorges University (Registry Identifier: China Three Gorges University)
Record Dates: First submitted 2014-03-24; First posted 2014-04-03 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Anesthesia
Keywords: intrathecal; ropivacaine; motor blockade; local anesthetics
MeSH Terms: interventions — Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- age: subjects stratified according to age: 20-30 years (Group 1), 31-40 years (Group 2), 41-50 years (Group 3), 51-60 years (Group 4), 61-70 years (Group 5), and 71-80 years (Group 6).
  Interventions: Other: age

INTERVENTIONS:
Other: age — subjects stratified according to age: 20-30 years (Group 1), 31-40 years (Group 2), 41-50 years (Group 3), 51-60 years (Group 4), 61-70 years (Group 5), and 71-80 years (Group 6).

SUMMARY:
The primary aim of this study was to determine the median effective dose (ED50) for motor block of intrathecally-administered ropivacaine in adults (20-80 years), and to assess the effect of age on ED50 required for motor block.

DETAILED DESCRIPTION:
This study was performed in adult patients undergoing transurethral, urological or lower limb surgery under combined spinal and epidural anesthesia. Patients were stratified according to age: 20-30, 31-40, 41-50, 51-60, 61-70, and 71-80 years. The spinal component of the anesthetic was established by bolus administration of various up-and-down doses of 0.75% ropivacaine, determined by Dixon's method, with the first patient receiving 15 mg, and with testing intervals of 1.5 mg according to failure or success of the preceding patient's motor block. The degree of motor block after intrathecal administration of each dose was evaluated by the modified Bromage and Hip motor function score. The primary outcome was obtained by administration of the mean dosage that was determined from the midpoints of all independent pairs of patients involving a crossover from failure to success during 5 minutes after the spinal injection. The ED50 were estimated from the up-and-down sequences using the method of Dixon and Massey and logistic regression. Other endpoints were included on the basis of sensory block level, duration of motor blockade, hypotension, and vasopressor requirements.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who were undergoing transurethral, urological or lower limb surgery, primarily under the spinal anesthesia

Exclusion Criteria:

* Patients with diabetes, obesity, neuromuscular diseases, bleeding diathesis, hypersensitivity to amide local anesthetics, lumbar vertebrae abnormality, chronic back pain, or who were pregnant

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who were undergoing transurethral, urological or lower limb surgery, primarily under the spinal anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
the dose of intrathecal ropivacaine | at 5-min after administered ropivacaine

CONTACTS AND LOCATIONS:
Overall Officials: jun yang, PhD, Study Director — China Three Gorges University
Locations (1):
- China Three Gorges University, Yichang, Hubei, China

REFERENCES:
- [Background] Lee YY, Ngan Kee WD, Fong SY, Liu JT, Gin T. The median effective dose of bupivacaine, levobupivacaine, and ropivacaine after intrathecal injection in lower limb surgery. Anesth Analg. 2009 Oct;109(4):1331-4. doi: 10.1213/ane.0b013e3181b1912b. PMID 19762766
- [Background] Gupta R, Bogra J, Singh PK, Saxena S, Chandra G, Kushwaha JK. Comparative study of intrathecal hyperbaric versus isobaric ropivacaine: A randomized control trial. Saudi J Anaesth. 2013 Jul;7(3):249-53. doi: 10.4103/1658-354X.115326. PMID 24015125